CLINICAL TRIAL: NCT05772650
Title: Healthier Together Mood Booster Challenge
Brief Title: The Online Mood Booster Challenge to Support Physical and Mental Health
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: McGill University (Other)
Responsible Party: Principal Investigator, Steven Grover, MD, Professor of Medicine, McGill University, McGill University
Other Study IDs: CLIN1903
Record Dates: First submitted 2023-02-13; First posted 2023-03-16 (Actual); Last update posted 2023-03-16 (Actual); Status verified 2023-03

CONDITIONS: Mental Health Wellness 1
Keywords: web based health promotion

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Behavioral: e-Health Program — Lifestyle modification for health and disease management using digital solutions

SUMMARY:
Healthier Together Mood Booster Challenge - To improve mental and physical fitness, while providing participants with online education, tracking, social connectivity, and feedback.

DETAILED DESCRIPTION:
An 8-week web-based health promotion program to learn strategies and use digital tools that will give participants a physical, mental, and emotional boost, with exercise remaining a key component of the mission.

Each week participants will learn and practice evidence-based strategies that they will master to improve their physical and mental health.

Techniques will be focused on: spending time exercising outdoors, practicing daily gratitude, practicing good posture, building social connection, deep breathing, listening to music, limiting time on social media and focusing on better sleep.

ELIGIBILITY:
Inclusion Criteria:

* Affiliated with McGill University or family member

Exclusion Criteria: None

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: McGill University faculty, staff, students and invited family members
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2023-02-06 (Actual); Primary Completion 2023-04-16 (Estimated); Study Completion 2023-06-30 (Estimated)

PRIMARY OUTCOMES:
Improvement in Physical Activity Levels | Feb 20 - April 16, 2023
  8 week program to create healthy habits of incorporating increased physical activity in daily life.
  Self-reported physical activity levels using the International Physical Activity Questionnaire (IPAQ) (weekly metabolic equivalents (METs); using an estimate of 4 METs/ min moderate exercise and 8 METs/ min vigorous exercise)
Adherence to Program | Feb 20 - April 16, 2023
  8 Week program to help change behaviour for healthy habit creation. Adherence will be measured as the number of days tracking physical activity levels and answering the behaviour change questions.
  Less than 7 days = very poor adherence 7-21 days = poor adherence 22-42 days = moderate adherence 43-49 days = good adherence Greater than 49 days = excellent adherence
Improvement in Stress | Feb 20 - April 16, 2023
  The following methodology will be used to measure the above metric:
  - Stress score - Perceived Stress Scale. 10 questions; Total score from 0 to 40; ≥18 high stress (1 standard deviation above the mean)
Improvement in Sleep | Feb 20 - April 16, 2023
  The following methodology will be used to measure the above metric:
  - Sleep score - Insomnia Severity Index. 7 questions; Total score from 0 to 28; ≥ 8 subthreshold insomnia
Improvement in Mood | Feb 20 - April 16, 2023
  The following methodology will be used to measure the above metric:
  - Depression score - Centre for Epidemiological Studies - Depression questionnaire 20 questions; Total score 0-40; ≥16 subthreshold depressive symptoms
Improvement in Burnout | Feb 20 - April 16, 2023
  The following methodology will be used to measure the above metric:
  - Burnout - Oldenburg burnout assessment. <2.89 no or little sign of burnout; 2.89 to 3.51 may be at risk of burnout; >3.51 at very high risk of burnout

CONTACTS AND LOCATIONS:
Overall Officials: Dr. Steven Grover, MD, Principal Investigator — McGill University
Locations (1):
- McGill University, Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: Undecided
Aggregate data analysis